CLINICAL TRIAL: NCT04496232
Title: Strategies for Reducing Sperm DNA Fragmentation in ICSI Semen Samples: a Prospective Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ganin Fertility Center (Other)
Responsible Party: Principal Investigator, Eman Hasanen, BSc., Ganin Fertility Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GFC-004
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Male Infertility
Keywords: Sperm DNA fragmentation; Second ejaculate; Sperm Selection; PICSI
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal SDF (No Intervention): Using routine semen processing method
- Physiological ICSI (PICSI) (Active Comparator): Sperm selection using PICSI dishes for selecting sperm with lower DNA fragmentation index for ICSI
  Interventions: Device: PICSI
- Second ejaculate (Active Comparator): Using the second ejaculate as a way of reducing SDF in the semen sample used for ICSI
  Interventions: Other: Second ejaculate

INTERVENTIONS:
Device: PICSI — Semen processing by density gradient centrifugation followed by sperm selection by PICSI dishes of the first ejaculate
  Arms: Physiological ICSI (PICSI)
Other: Second ejaculate — Semen processing by density gradient centrifugation for the second ejaculate
  Arms: Second ejaculate

SUMMARY:
Comparing second ejaculate and physiological ICSI (PICSI) as strategies for improvement of abnormal sperm DNA fragmentation in patients undergoing ICSI.

DETAILED DESCRIPTION:
Sperm DNA fragmentation has shown a negative correlation with embryo quality, fertilization, implantation, clinical pregnancy, and live birth rates. And a positive correlation with the miscarriage rate. Abnormal sperm DNA fragmentation can be improved through the second ejaculate strategy, by limiting the time of sperm presence in the epididymis. PICSI is a robust sperm selection technique that can select individual mature intact sperm DNA. In our study, we will compare PICSI as a valid sperm selection technique to second ejaculate, as a natural cost-free strategy to manage abnormal SDF. In addition to a normal SDF arm as a control.

ELIGIBILITY:
Inclusion Criteria:

* Male partner with abnormal sperm DNA fragmentation index (>20%) by TUNEL assay
* Male partner with at least 1 million progressive motile count
* Male aged 18-50 years
* Male with adjusted sexual abstinence days (1-2 days)
* Female aged 18-37 years
* Normo-responder females (at least 5 mature oocytes)

Exclusion Criteria:

* Leukocytospermia
* Varicocele
* Known genetic abnormality
* Use of oocyte or sperm donors
* Use of a gestational carrier
* Presence of any endometrial factors that can affect embryo implantation
* Any contradictions to undergoing in vitro fertilization or gonadotropin stimulation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Fertilization rate | 16-19 hours
  Defined as the proportion of fertilized oocytes over the injected oocytes.
Cleavage rate | 3 days
  Defined as the proportion of cleaved embryos on day 3 over the injected oocytes.
Blastulation rate | 5-6 days
  Defined as the proportion of blastocysts formed on day 5 or 6 over the cleaved embryos on day 3.
Blastocyst quality rate | 5-6 days
  Defined as the assessment of blastocyst quality according to Gardner's criteria into: good, fair, or bad in terms of percentage of the total formed blastocysts.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Hasanen, Principal Investigator — Ganin Fertility Center; Radwa Omar, Principal Investigator — Ganin Fertility Center; Hanaa Alkhader, Principal Investigator — Ganin Fertility Center; Hosam Zaki, MSc, FRCOG, Study Director — Ganin Fertility Center; Manar Hozayen, MSc., Principal Investigator — Ganin Fertility Center
Locations (1):
- Ganin Fertility Center, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP